CLINICAL TRIAL: NCT01772446
Title: Effectiveness of Sending Sms Text Messages to Mobile Phone Patients to Remind Upcoming Appointments and Improve the Control of Diabetic Patients in Primary Care
Brief Title: Effectiveness of SMS in Diabetes Control
Acronym: SMSaludD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Raquel Cobos Campos, Epidemiologist, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PAPPS-01
Record Dates: First submitted 2013-01-10; First posted 2013-01-21 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes
Keywords: diabetes; management; glycated hemoglobin; preventive activities
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL GROUP (No Intervention): ROUTINE CLINICAL PRACTICE
- SMS MESSAGING (Experimental): SMS MESSAGES TO MOBILE PHONE TO REMEMBER THE NEXT CONTROL OF GLYCATED HEMOGLOBIN
  Interventions: Behavioral: SMS MESSAGING

INTERVENTIONS:
Behavioral: SMS MESSAGING — SMS MESSAGING TO MOBILE PHONE TO REMEMBER THE NEXT CONTROL OF GLYCATED DIABETES
  Arms: SMS MESSAGING

SUMMARY:
Introduction: The Spanish Society of Family and Community Medicine, started the Program of Preventive Activities and Health Promotion, which generates periodic recommendations of preventive methods based on scientific evidence. In the last update it has become evident the need of modifications to adapt the program to modern times and focuses on improving accessibility and offering more flexible responses to users of the program. In this sense, the mobile phone technology could be useful, specifically the messaging service to remind patients their appointments and increase attendance rates. Main objective Compare the percentage of patients in the intervention group compared with the control group who achieved a figure of HbA1c <7% in 2013.Design: single blind Randomized Clinical Trial. Study population: Patients with diabetes with or without hypertension or lipid metabolism disorder, over 18 years, belonging to the Public Health System of Basque Country (primary care) meeting the inclusion / exclusion criteria. Sample size: 238 patients (119 per arm) to detect a difference of 16% in the percentage of patients with HbA1c lower than 7% between groups: Short Messages Standard (SMS) group: Mobile messages reminding the next review of Papps. Control group: Routine clinical practice. Statistical analysis: The relationship between the intervention received and the main variable (compliance with preventive activities at 12 months) were analyzed using a logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with or without hypertension or lipid metabolism disorder,
* Aged between 35 and 74 years old with or without hypertension or lipid metabolism disorder,
* Mobile phone holder,
* Able to read messages via mobile phone.

Exclusion criteria:

* Pregnant women,
* Patients whose next date for HbA1c control is less than 2 months
* Patients with HbA1c <7%

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compare the percentage of patients in the intervention group versus the control group who get a HbA1c below 7% | 12 months

SECONDARY OUTCOMES:
Compare the mean change in HbA1c values between SMS group patients and control patients | 6 and 12 months
Compare the percentage of patients in the intervention group compared with the control group that meet the following preventive recommendations | 12 months
In patients with predictive risk index <1.5, to compare the incidence of diabetic complications in each group | 12 months
Evaluate the percentage of patients who are controlled. We consider controlled patient when HbA1C <7%, BP <140/80 and cardiovascular risk <20% measured by the scale of Heart Register of Gerona (REGICOR) | 6 and 12 months
To identify factors associated with better compliance of preventive activities in both groups | 12 months
Evaluate whether the intervention is more effective (reducing HbA1c below 7%) in patients with predictive risk index <1.5, or in patients with predictive risk index> 1.5. | at 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Comarca Araba, Vitoria-Gasteiz, Álava, Spain